CLINICAL TRIAL: NCT01585844
Title: Obstructive Sleep Apnea in Pregnancy:Epidemiology and Maternal/ Neonatal Morbidity
Brief Title: Sleep Apnea in Pregnancy Screening Study
Acronym: SAPSS
Status: Completed | Type: Observational
Sponsor: MetroHealth Medical Center (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: RWJ64323
Record Dates: First submitted 2012-04-23; First posted 2012-04-26 (Estimated); Last update posted 2023-11-14 (Actual); Status verified 2012-04

CONDITIONS: Sleep Apnea; Obesity
Keywords: sleep apnea; pregnancy; obesity
MeSH Terms: conditions — Sleep Apnea Syndromes; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Women with sleep apnea
- Women without sleep apnea

SUMMARY:
Obstructive sleep apnea is known to be a significant source of morbidity in the general population. It has been proposed to be associated with the development of preeclampsia and fetal growth restriction. As these are conditions that have long term maternal and neonatal implications, further information may help improve maternal/fetal outcome. One reason why women and in particular pregnant women are under diagnosed is the lack of an effective, reliable screening tool. Validated questionnaires used in the general population may not be effective in screening pregnant women. The investigators hypothesize that sleep apnea will have 20% prevalence in the obese pregnant population and that it is associated with increased maternal and neonatal morbidity. The investigators will recruit obese pregnant women in their prenatal care clinics and they will be screened for OSA using validated sleep questionnaires including the Epworth sleepiness scale, the Fatigue Scale and the Berlin Questionnaire. The subjects will then perform overnight apnea monitoring utilizing a portable sleep apnea detection device. Women who meet clinical criteria for OSA will be referred for overnight polysomnogram and management by the Pulmonary and Critical Care Division of the Internal Medicine Department. For all enrolled patients the remainder of prenatal care will be per routine. Data will be collected regarding the pregnancy course and outcomes.

The primary outcome of interest is the prevalence of sleep apnea in obese women and the associated maternal and neonatal morbidity. The secondary outcome measures will be molecular measures of systemic inflammation, oxidative stress and angiogenesis associated with sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* Prepregnancy BMI of 30kg/m2 or greater
* Singleton pregnancy
* 18 years or older

Exclusion Criteria:

* Chronic use of narcotics or other CNS drugs
* Inability to sleep beyond 2 hours
* 3 or more missed prenatal visits

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Obstetric care clinic at a tertiary care hospital
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2008-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
The prevalence of sleep apnea in obese pregnant women | Subjects will be followed for the duration of their pregnancy and postpartum period, an expected average of 26 weeks

SECONDARY OUTCOMES:
Alterations in biomarkers of inflammation and oxidative stress | Subjects will be followed for the duration of their pregnancy and postpartum period, an expected average of 26 weeks
The prevalence of maternal and neonatal morbidity | Subjects will be followed for the duration of their pregnancy and postpartum period, an expected average of 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Judette Louis, MD, MPH, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Connolly G, Razak AR, Hayanga A, Russell A, McKenna P, McNicholas WT. Inspiratory flow limitation during sleep in pre-eclampsia: comparison with normal pregnant and nonpregnant women. Eur Respir J. 2001 Oct;18(4):672-6. doi: 10.1183/09031936.01.00053501. PMID 11716173
- [Background] Young T, Peppard PE, Gottlieb DJ. Epidemiology of obstructive sleep apnea: a population health perspective. Am J Respir Crit Care Med. 2002 May 1;165(9):1217-39. doi: 10.1164/rccm.2109080. PMID 11991871
- [Background] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434
- [Background] Joel-Cohen SJ, Schoenfeld A. Fetal response to periodic sleep apnea: a new syndrome in obstetrics. Eur J Obstet Gynecol Reprod Biol. 1978 Apr;8(2):77-81. doi: 10.1016/0028-2243(78)90131-4. PMID 45501
- [Background] Franklin KA, Holmgren PA, Jonsson F, Poromaa N, Stenlund H, Svanborg E. Snoring, pregnancy-induced hypertension, and growth retardation of the fetus. Chest. 2000 Jan;117(1):137-41. doi: 10.1378/chest.117.1.137. PMID 10631211
- [Background] Charbonneau M, Falcone T, Cosio MG, Levy RD. Obstructive sleep apnea during pregnancy. Therapy and implications for fetal health. Am Rev Respir Dis. 1991 Aug;144(2):461-3. doi: 10.1164/ajrccm/144.2.461. PMID 1859076
- [Background] Louis JM, Auckley D, Sokol RJ, Mercer BM. Maternal and neonatal morbidities associated with obstructive sleep apnea complicating pregnancy. Am J Obstet Gynecol. 2010 Mar;202(3):261.e1-5. doi: 10.1016/j.ajog.2009.10.867. Epub 2009 Dec 14. PMID 20005507
- [Background] Pien GW, Fife D, Pack AI, Nkwuo JE, Schwab RJ. Changes in symptoms of sleep-disordered breathing during pregnancy. Sleep. 2005 Oct;28(10):1299-305. doi: 10.1093/sleep/28.10.1299. PMID 16295215